CLINICAL TRIAL: NCT01253967
Title: Hospital-based Surveillance to Estimate the Disease Burden of Rotavirus Gastroenteritis in Children < 5 Years of Age in Romania
Brief Title: Surveillance Study to Estimate the Proportion of Rotavirus Gastroenteritis in Children < 5 Years of Age in Romania
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 110436
Record Dates: First submitted 2010-11-30; First posted 2010-12-06 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Rotavirus
Keywords: Gastroenteritis; Hospital surveillance; Rotavirus gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples

GROUPS / COHORTS (3):
- Group A: Subjects who are hospitalised for acute gastroenteritis
  Interventions: Procedure: Collection of stool samples; Other: Health economics questionnaire
- Group B: Subjects who visit an emergency room for acute gastroenteritis
  Interventions: Procedure: Collection of stool samples; Other: Health economics questionnaire
- Group C: Subjects who have rotavirus positive laboratory results and developed acute gastroenteritis at least 48 hours after hospitalisation.
  Interventions: Procedure: Collection of stool samples; Other: Health economics questionnaire

INTERVENTIONS:
Procedure: Collection of stool samples — Stool samples will be tested for the presence of rotavirus and a subset of rotavirus positive samples will be genotyped.
Other: Health economics questionnaire — For a subset of subjects, additional economic data will be gathered by completing a questionnaire

SUMMARY:
The purpose of this hospital based study is to estimate the proportion of rotavirus gastroenteritis in children < 5 years of age in Romania.

DETAILED DESCRIPTION:
The study consist of a main study and a health economics study

Main study: The study will focus on three different groups of patients:

* Subjects who are hospitalised for acute gastroenteritis.
* Subjects who visit an emergency room for acute gastroenteritis.
* Subjects who have rotavirus positive laboratory results and developed acute gastroenteritis at least 48 hours after hospitalisation.

Health economics study: for a subset of subjects, additional economic data will be gathered by completing a questionnaire

ELIGIBILITY:
Inclusion Criteria:

* A male or female child aged < 5 years at the time of admission. A child becomes ineligible on the day of her/his fifth birthday.
* A subject, who during the study period:

  * Is hospitalised for acute gastroenteritis Or
  * Visits an emergency room for acute gastroenteritis Or
  * Has rotavirus positive laboratory results and develops acute gastroenteritis at least 48 hours after hospitalisation

Exclusion Criteria:

Not applicable

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 5 years of age treated at a hospital site (subjects hospitalised with community acquired acute gastroenteritis, subjects who visited the emergency room for acute gastroenteritis or subjects with medical care associated rotavirus infection).
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of rotavirus gastroenteritis among all acute gastroenteritis hospitalisations of children < 5 years of age | At least 12 months from study start
Proportion of rotavirus gastroenteritis among all acute gastroenteritis emergency room visits for children < 5 years of age | At least 12 months from study start
Incidence of medical care associated rotavirus gastroenteritis among all hospitalised children < 5 years of age | At least 12 months from study start

SECONDARY OUTCOMES:
Age distribution of children with rotavirus gastroenteritis | At least 12 months from study start
Percentage of rotavirus genotypes amongst all isolated strains in children < 5 years of age | At least 12 months from study start
Potential risk factors for rotavirus gastroenteritis | At least 12 months from study start
Rotavirus gastroenteritis associated costs | At least 12 months from study start
Proportion of acute gastroenteritis among all hospitalisations of children < 5 years of age | At least 12 months from study start
Proportion of community acquired acute gastroenteritis among all emergency room visits for children < 5 years of age | At least 12 months from study start
Seasonal distribution (if appropriate) of rotavirus among all children < 5 years of age | At least 12 months from study start
Severity of rotavirus among all children < 5 years of age | At least 12 months from study
Proportion of rotavirus gastroenteritis among all hospitalisations of children < 5 years of age | At least 12 months from study start
Proportion of community acquired rotavirus gastroenteritis among all emergency room visits for children < 5 years of age | At least 12 months from study start

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Sibiu
  - GSK Investigational Site, Timișoara

REFERENCES:
- [Derived] Benea OE, Streinu-Cercel A, Dorobat C, Rugina S, Negrutiu L, Cupsa A, Duiculescu D, Chiriac C, Itu C, Prisacariu LJ, Iosif I. Efficacy and safety of darunavir (Prezista((R))) with low-dose ritonavir and other antiretroviral medications in subtype F HIV-1 infected, treatment-experienced subjects in Romania: a post-authorization, open-label, one-cohort, non-interventional, prospective study. Germs. 2014 Sep 1;4(3):59-69. doi: 10.11599/germs.2014.1057. eCollection 2014 Sep. PMID 25276665
- [Derived] Anca IA, Furtunescu FL, Plesca D, Streinu-Cercel A, Rugina S, Holl K. Hospital-based surveillance to estimate the burden of rotavirus gastroenteritis in children below five years of age in Romania. Germs. 2014 Jun 2;4(2):30-40. doi: 10.11599/germs.2014.1053. eCollection 2014 Jun. PMID 24967217